CLINICAL TRIAL: NCT01119079
Title: A Randomized, Prospective Study to Establish Whether the Instillation of 10ml of Epidural Normal Saline Improves the Quality Of Epidural Analgesia During Labor
Brief Title: Study to Determine Whether the Instillation of 10ml Normal Saline Improves Epidural Analgesia During Labor
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: PI unable to recruit appropriate patients
Sponsor: University of Medicine and Dentistry of New Jersey (Other)
Responsible Party: Sponsor
Organization: Rutgers, The State University of New Jersey (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0120090228
Record Dates: First submitted 2010-05-06; First posted 2010-05-07 (Estimated); Last update posted 2015-04-24 (Estimated); Status verified 2015-04

CONDITIONS: Parturients
Keywords: labor pain; epidural
MeSH Terms: conditions — Labor Pain | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard labor epidural protocol (Placebo Comparator): Standard labor epidural protocol
  Interventions: Procedure: Administration of epidural anesthesia for labor
- 10ml Normal Saline prior to lidocaine (Experimental)
  Interventions: Other: Normal Saline

INTERVENTIONS:
Other: Normal Saline — 10ml Normal Saline instilled in the epidural space
  Arms: 10ml Normal Saline prior to lidocaine
Procedure: Administration of epidural anesthesia for labor — Standard procedure
  Arms: Standard labor epidural protocol

SUMMARY:
In current obstetric anesthesia practice, epidural analgesia is the most effective technique to control labor pain for those women who request pain-free delivery. Epidural analgesia not only allows us to obtain greater pain relief and increased satisfaction of mothers, but also permits us to convert it to regional anesthesia in case of operative delivery, avoiding general anesthesia.

One of the major concerns with epidural anesthesia in labor setting is the inability to produce an intensive analgesia or adequate level to proceed with cesarean section. This study is designed to examine the hypothesis that 10ml epidural normal saline to reduce rate of one-side block, low segmental block, and patch block, and improve quality of labor epidural analgesia/ anesthesia in obstetric population.

DETAILED DESCRIPTION:
One of the major concerns with epidural anesthesia in labor setting is the inability to produce an intensive analgesia or adequate level to proceed with cesarean section. The incidence of this event is rather various among reports, reflecting variability in definitions, authors' clinical judgment and perception, practice parameters, hospital settings. In most of related studies, the term of incomplete block was used and defined as (1) unilateral block; (2) unblocked sacral segments; (3) low level; (4) unblocked segments or a patchy block. 1Reported incidence of inadequate analgesia/anesthesia was 18% to 31.8%. In addition, the reported incidence of intraoperative discomfort/visceral pain was from 10% to 56%.1

If the anesthesia/analgesia is not adequate, other treatment modalities have to be provided to improve pain relief, these include intravenous narcotics or ketamine, replacements of epidural catheter, or general anesthesia, the risks of complications may be increased by those managements.

The etiology and mechanisms of failed or dysfunctional epidural analgesia or anesthesia in obstetrics are complex, multifactorial, and not entirely understood. Depending on the situation, the causes might be evident or puzzling and difficult to explain.

Injection of fluid is frequently used for identification of the epidural space by the loss-of-resistance (LOR) technique. It has been shown that different volumes of saline may affect the subsequent epidural analgesia. Iwama showed that using 10 mL of saline as compared to two mL in patients undergoing elective surgery during lumbar epidural anesthesia with 2% mepivacaine resulted in a greater extent of anesthesia.2 Also, Okutomi et al examined the effect of saline volume on anesthetic levels and quality of thoracic epidural block in patients undergoing upper abdominal surgery. They demonstrated that the block level for cold after mepivacaine 1.5% was proportional to the saline volume injected, whereas the block level for pain was independent of the saline solution.3 Identifying the epidural space by a lost of resistance to air method is thought to increase the incidence of inadequate anesthesia. A randomized study, comparing air versus saline to identify the epidural space in parturients, found a higher incidence of inadequate analgesia in the air group (36% versus 19%).4

In parturients requesting epidural analgesia, a few studies showed that 2- 10ml normal saline giving to epidural space after LOR was obtained reduced the rate of venous puncture and unblock segments to cold and pin prick, but did not improve the visual analog pain scale or reduced the need for supplemental.3,5,6 No study on improvement of unilateral block, patch block and patients' satisfaction in obstetric setting has been found.

We design this study to examine the hypothesis that 10ml epidural normal saline to reduce rate of one-side block, low segmental block, and patch block, and improve quality of labor epidural analgesia/ anesthesia in obstetric population.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists class I-II term parturients with singleton vertex presentation in active labor
* Patients who have cervical dilatation between 3 and 7 centimeters

Exclusion Criteria:

* • Patients with contraindications to epidural analgesia,

  * severe medical or obstetric complications,
  * morbid obesity (body mass index >40 kg/m2),
  * history of drug or alcohol abuse,
  * abnormal hepatic (AST/ALT), renal (creatinine levels), or hematological (PTT levels) test results.
  * presence of blood on the second insertion into the intervertebral space
  * presence of cerebral spinal fluid upon insertion into the intervertebral space
  * subjects who deliver (either vaginally or via cesarean section) within 2 hours of the epidural insertion
  * subjects less than 36 weeks gestation

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2010-03; Primary Completion 2012-06 (Estimated); Study Completion 2012-09 (Estimated)

PRIMARY OUTCOMES:
improve quality of labor epidural analgesia/ anesthesia in obstetric population. | Administration of epidural anesthesia + 2 hours

CONTACTS AND LOCATIONS:
Overall Officials: Dongchen Li, MD, PhD, Principal Investigator — UMDNJ-NJMS
Locations (1):
- University Hospital, Newark, New Jersey, United States